CLINICAL TRIAL: NCT05792540
Title: Clinical Study to Evaluate the Possible Efficacy of Dapagliflozin and Atorvastatin in Patients With Major Depressive Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Manal Ali Mahrous Hamouda Faculty of Pharmacy, Menufia University (Unknown)
Responsible Party: Principal Investigator, Mostafa Bahaa, Teaching Assistant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4/2023
Record Dates: First submitted 2023-03-19; First posted 2023-03-31 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Fluoxetine; dapagliflozin; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Control group ( fluoxetine 20 mg, n =25 ) who will receive fluoxetine (20 mg) once daily for 3 months
  Interventions: Drug: Fluoxetine 20 mg
- Dapagliflozin group (Active Comparator): Patients will receive fluoxetine (20 mg) once daily plus dapagliflozin 10 mg once daily for 3 months
  Interventions: Drug: Fluoxetine 20 mg; Drug: Dapagliflozin 10mg Tab
- Atorvastatin group (Active Comparator): Patients will receive fluoxetine (20 mg) once daily plus atorvastatin 80 mg once daily for 3 months
  Interventions: Drug: Fluoxetine 20 mg; Drug: Atorvastatin 80mg

INTERVENTIONS:
Drug: Fluoxetine 20 mg — Fluoxetine is a type of antidepressant known as a selective serotonin reuptake inhibitor (SSRI). It's often used to treat depression, and sometimes obsessive-compulsive disorder and bulimia. It works by increasing the levels of serotonin in the brain
Drug: Dapagliflozin 10mg Tab — Dapagliflozin (DAPA), a sodium-glucose co-transporter 2 inhibitor (SGLT2-I), has proven to be an effective hyperglycemic suppressor due to its role in inhibiting the reabsorption of 30-50% of the glucose filtered by the kidney, besides its role in the improvement of insulin resistance
  Arms: Dapagliflozin group
Drug: Atorvastatin 80mg — Atorvastatin is a synthetic and lipophilic statin, a class of drugs used in the treatment of hypercholesterolemia
  Arms: Atorvastatin group

SUMMARY:
Major depressive disorder (MDD) is a significant cause of disability that affects approximately 16% of the world's population and is associated with chronic inflammation. Although the mechanisms of MDD have not yet been clearly elucidated, NLRP3 inflammasomes have been implicated in the pathogenesis of depression.NLRP3 inflammasome is an intracellular multiprotein complex that consists of nod-like receptor protein 3, an adaptor protein, and a procaspase-1 precursor. It is well known that a variety of danger signals, such as pathogen-associated molecular patterns and danger-associated molecular patterns can activate NLRP3 inflammasome

ELIGIBILITY:
Inclusion Criteria:

- Age ≥ 18 years Both males and females will be included Negative pregnancy test and effective contraception. Depressed patients for at least 2 months with a Hamilton rating score of more than 18.

Exclusion Criteria:

* Patients with bipolar I or bipolar II disorder
* Patients with personality disorders
* Patients with eating disorders
* Patients with substance dependence or abuse
* Patients with concurrent active medical conditions
* Patients with a history of seizures
* Patients with a history of receiving Electroconvulsive therapy (ECT)
* Patients with inflammatory disorders
* Patients with allergies or contraindications to the used medications
* Patients with finally pregnant or lactating females
* Diabetic or hyperlipidaemic patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
• The primary endpoint is the change in Hamilton Rating Scale | 3 months
  • The primary endpoint is the change in Hamilton Rating Scale

SECONDARY OUTCOMES:
The secondary endpoint is estimated by changes in serum biomarkers. | 3 months
  The secondary endpoint is estimated by changes in serum biomarkers such as F) Nuclear factor erythroid 2-related factor 2

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Menoufia University, Tanta, Shebeen El-Kom, Egypt

REFERENCES:
- [Derived] Aldossary KM, Ali LS, Abdallah MS, Bahaa MM, Elmasry TA, Elberri EI, Kotkata FA, El Sabaa RM, Elmorsi YM, Kamel MM, Negm WA, Elberri AI, Hamouda AO, AlRasheed HA, Salahuddin MM, Yasser M, Hamouda MA. Effect of a high dose atorvastatin as added-on therapy on symptoms and serum AMPK/NLRP3 inflammasome and IL-6/STAT3 axes in patients with major depressive disorder: randomized controlled clinical study. Front Pharmacol. 2024 May 24;15:1381523. doi: 10.3389/fphar.2024.1381523. eCollection 2024. PMID 38855751